CLINICAL TRIAL: NCT05840029
Title: THE ROLE OF VIDEO-ASSISTED THORACOSCOPIC SURGERY IN PATIENTS WITH ADVANCED OVARIAN MALIGNANCIES
Brief Title: VATS IN PATIENTS WITH ADVANCED OVARIAN MALIGNANCIES
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Other Study IDs: VATS and ovarian cancer
Record Dates: First submitted 2023-04-21; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2022-11

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer stage III, IV; VATS, CT staging
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Patients who will get neoadjuvant chemotherapy based on VATS finding.: Patients will be considered to receive neoadjuvant chemotherapy if there is residual intrathoracic disease
  Interventions: Procedure: VIDEO-ASSISTED THORACOSCOPIC SURGERY
- Group B: Patients who will proceed into debulking surgery based on VATS finding.: Patients will be considered to be eligible for complete debulking, if VATS showed no intrathoracic tumor or if VATS achieves complete removal of tumor nodules through intraoperative frozen section histopathological examination.
  Interventions: Procedure: VIDEO-ASSISTED THORACOSCOPIC SURGERY

INTERVENTIONS:
Procedure: VIDEO-ASSISTED THORACOSCOPIC SURGERY — A minimally invasive approach, to not only drain the pleural effusion but also evaluate macroscopic pleural disease and, when possible, resect gross tumor.
  Other Names: VATS

SUMMARY:
Ovarian cancer is the seventh most common cancer and the fifth leading cause of death in women worldwide.

About 70% of patients with epithelial ovarian cancer present with advanced disease which will require a combination of cytoreductive surgery and chemotherapy to give them their best chance of long term survival.The presence of macroscopic pleural disease-especially if undetected and unresected after primary debulking surgery-may alter treatment decision-making and markedly affect survival. Video-Assisted Thoracoscopic Surgery (VATS) allows surgeons, through a minimally invasive approach, to not only drain the pleural effusion but also evaluate macroscopic pleural disease and, when possible, resect gross tumor.

Few studies reported that VATS altered the therapeutic management in ovarian cancer patients leading to an upstaging or down-staging when compared to the CT staging. Therefore, this study will prospectively assess the role of VATS in the diagnosis and management of supradiaphragmatic disease as well as evaluate the impact of VATS findings on the decision of surgical management in patients with advanced ovarian cancer FIGO (The International Federation of Gynecology and Obstetrics) stage III/IV.

ELIGIBILITY:
Inclusion Criteria:

* FIGO stage III/IV ovarian cancer with or without pleural effusion

Exclusion Criteria:

1. Previously treated ovarian disease.
2. Patient unfit for single lung ventilation.
3. Patients with previous lung surgery.
4. Patients with possible intrapleural adhesions.
5. Patients who had pulmonary resection.

Ages: 20 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients with advanced ovarian cancer at gyneoncology department will be enrolled
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Prediction of intrathoracic disease using chest-CT results compared to the standard reference results using VATs | 3 weekS
  Comparison between the Chest-CT results in preoperative evaluation of supra-diaphragmatic disease will be compared to the intra-operative VATS evaluation results to evaluate the role of the VATS in those patients

SECONDARY OUTCOMES:
The rate of change in the treatment plan according to VATs results | 1 week
  The number of patients that will receive different treatment plan after detection of intrathoracic disease using VATs

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University, Alexandria, Egypt